CLINICAL TRIAL: NCT00142922
Title: Breaking Down Barriers to Diabetes Self-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DK 60115 (completed); DK 60115; CHS00-34
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Adherence; self-care; Behavioral intervention; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Attended Breaking Down Barriers program
  Interventions: Behavioral: Breaking Down Barriers
- 2 (Active Comparator): Attention control group
  Interventions: Behavioral: Breaking Down Barriers
- 3 (Active Comparator): Indivdual attention control group
  Interventions: Behavioral: Breaking Down Barriers

INTERVENTIONS:
Behavioral: Breaking Down Barriers — completed

SUMMARY:
Performance of self-care recommendations is key to the successful treatment of diabetes. However, many patients have difficulty adhering to diabetes self-care recommendations. Recent results from our own studies and others have identified specific barriers to diabetes self-care. To evaluate the efficacy of a diabetes educator-led group intervention, the Breaking Down Barriers Program, that addresses barriers and therefore leads to improved adherence to diabetes self-care recommendations, we will randomize 222 (111 type 1 and 111 type 2) diabetes patients to one of three conditions: 1) the Breaking Down Barriers Program, 2) a cholesterol attention control condition, or 3) a 'usual care' control condition. We hypothesize that those assigned to the Breaking Down Barriers group will improve self-care behaviors and glycemic control more than those in the two control groups. We will follow study subjects for one year to determine whether their self-care behaviors and glycemic control improved and if the improvement was maintained over time.

ELIGIBILITY:
Inclusion Criteria:

For Patients With Type 1 Diabetes

* Aged 18-65
* Presence of type 1 diabetes mellitus.
* 2-25 year duration.

For Patients With Type 2 Diabetes

* Aged 25-65 years
* presence of type 2 diabetes mellitus.
* 2 years since initial diagnosis.

Exclusion Criteria:

* Renal disease, microalbumin >300 ug/mg)
* Severe peripheral diabetic neuropathy and/or severe peripheral vascular disease
* Symptomatic severe autonomic neuropathy who may be at risk when increasing activity levels.
* Women who are currently pregnant
* proliferative diabetic retinopathy based on dilated eye examination within one year of study entry. Patients whose eye disease is successfully treated will be included.
* HbA1c levels less than 7.0% (normal range 4.0 - 6.0%).
* HbA1c levels greater than 14.0%
* patients who underwent intensive insulin treatment within one year
* a history of severe, unstable myocardial infarction, congestive heart failure or other severe cardiac disease, severe hypertension (systolic more than 160 mmHg or diastolic 90 mmHg) who may be at risk when mildly increasing physical activity
* a DSMIV diagnosis of eating disorders including anorexia nervosa, bulimia, and severe weight-related insulin omission.
* Patients with recent diagnosis (past 6 months) of bipolar disorder, schizophrenia, mental retardation, organic mental disorder, and alcohol or drug abuse
* Patients whose diabetes diagnosed cannot be clearly classified as type 1 or type 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222
Dates: Start 2002-10; Study Completion 2007-10

PRIMARY OUTCOMES:
Self-Care Behaviors
Glycemic control (HbA1c)
fitness

SECONDARY OUTCOMES:
Quality of life
Diabetes Related emaitonal distress

CONTACTS AND LOCATIONS:
Overall Officials: Katie Weinger, EdD, Principal Investigator — Joslin Diabetes Center/Harvard Medical School
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Weinger K, Beverly EA, Lee Y, Sitnokov L, Ganda OP, Caballero AE. The effect of a structured behavioral intervention on poorly controlled diabetes: a randomized controlled trial. Arch Intern Med. 2011 Dec 12;171(22):1990-9. doi: 10.1001/archinternmed.2011.502. Epub 2011 Oct 10. PMID 21986346